CLINICAL TRIAL: NCT00005633
Title: Vaccination of Melanoma Patients With Tyrosinase YMD and gp100 IMD-Javelin Fusion Peptides/HSP70 Complexes: A Trial Comparing the Immunogenicity of Three Doses
Brief Title: Vaccine Therapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-036; CDR0000067788 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1771
Record Dates: First submitted 2000-05-02; First posted 2004-07-26 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — HSP70 Heat-Shock Proteins

INTERVENTIONS:
Biological: OVA BiP peptide
Biological: gp209-2M antigen
Biological: recombinant 70-kD heat-shock protein
Biological: tyrosinase peptide

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether active specific immunization comprising tyrosinase and gp100:209-217 (gp100) peptides fused with OVA BiP peptide and heat shock protein 70 (HSP70) induces immunity against tyrosinase and gp100 in HLA-A2 positive patients with stage III or IV melanoma. II. Determine the lowest optimally immunogenic dose of tyrosinase and gp100 in these patients. III. Determine the tolerability of this regimen in these patients.

OUTLINE: This is a dose escalation study of tyrosinase and gp100:209-217 antigen (gp100). Patients receive vaccination comprising tyrosinase and gp100 fused with OVA BiP peptide and heat shock protein 70 (HSP70) subcutaneously on weeks 0, 1, 2, 6, and 18 for a total of 5 vaccinations in the absence of disease progression or unacceptable toxicity. Cohorts of 9 patients receive escalating doses of tyrosinase and gp100 until the lowest optimally immunogenic dose is determined. The lowest optimally immunogenic dose is defined as the dose at which 4 or more of 9 patients demonstrate T-cell responses.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage III or IV melanoma that is in remission for 2-52 weeks after surgical resection OR minimally resectable HLA-A2 positive Patients who are candidates for potentially curative surgery not eligible until after surgery

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 80-100% Life expectancy: Not specified Hematopoietic: WBC greater than 3,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 2.5 mg/dL AST less than 74 Units/L LDH less than 400 Units/L Alkaline phosphatase no greater than 1.5 times upper limit of normal Renal: Not specified Pulmonary: No evidence of disease by chest x-ray or chest CT scan If pulmonary function tests are abnormal, then abdominal CT scan must be performed Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception No other high risk malignancy within the past 2 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No other medical condition that would preclude compliance or immunologic response No new metastasis during study that requires chemotherapy or radiotherapy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No concurrent chemotherapy Endocrine therapy: No corticosteroids during the interval between 1 week prior to each immunization through 2 weeks after each immunization Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: No antiinflammatory agents (e.g., aspirin) or other nonsteroidal antiinflammatory drugs during the interval between 1 week prior to each immunization through 2 weeks after each immunization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip O. Livingston, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States